CLINICAL TRIAL: NCT02300077
Title: Methadone in Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201408002
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Post-operative Pain; Anesthesia
Keywords: fentanyl, morphine; methadone
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Control (Intra-operative administration of opioids, other than methadone)
  Interventions: Drug: Control (Intra-operative administration of opioids, other than methadone)
- Treatment methadone 0.1 mg/kg (Active Comparator): methadone 0.1 mg/kg
  Interventions: Drug: methadone
- Treatment methadone 0.15 mg/kg (Active Comparator)
  Interventions: Drug: methadone

INTERVENTIONS:
Drug: methadone — Escalating dose of methadone up to .3mg/kg.
  Other Names: Dolophine
  Arms: Treatment methadone 0.1 mg/kg; Treatment methadone 0.15 mg/kg
Drug: Control (Intra-operative administration of opioids, other than methadone) — Intra-operative administration of opioids, other than methadone
  Other Names: morphine fentanyl
  Arms: Control

SUMMARY:
The μ-opioid receptor agonist methadone is frequently used in adult anesthesia and adult pain therapy. Methadone has an extremely long half-life, which confers therapeutic advantage by providing more stable plasma concentrations and long-lasting pain relief. Methadone perioperative pharmacokinetics and effectiveness in perioperative pain relief in inpatients is well characterized. There is, however, no information on methadone use in an ambulatory surgery setting and outpatient procedures. This pilot investigation will determine effectiveness of intraoperative methadone in reducing postoperative opioid consumption and providing improved pain relief in patients undergoing moderately painful, ambulatory surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Undergoing general anesthesia and moderately painful, ambulatory surgical procedures with anticipated overnight, postop hospital stay of < 24 hours
* Signed, written, informed consent

Exclusion Criteria:

* History of or known liver or kidney disease.
* Females who are pregnant or nursing.
* Opioid tolerant patients (e.g. preoperative methadone therapy or use of fentanyl transdermal patches)
* History of allergy to methadone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helga Komen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Komen H, Brunt LM, Deych E, Blood J, Kharasch ED. Intraoperative Methadone in Same-Day Ambulatory Surgery: A Randomized, Double-Blinded, Dose-Finding Pilot Study. Anesth Analg. 2019 Apr;128(4):802-810. doi: 10.1213/ANE.0000000000003464. PMID 29847382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done between March 2015-May 2016.
Pre-assignment Details: We withdrew 4 patients after consenting - two of patients met exclusion criteria, one patient withdrew consent, one anesthesia provider refused to participate the study.
Groups:
- Treatment Methadone 0.1 mg/kg: methadone
  methadone: Escalating dose of methadone up to .3mg/kg.
- Treatment Methadone 0.15 mg/kg: methadone
Period: Overall Study
Arm/Group | Control | Treatment Methadone 0.1 mg/kg | Treatment Methadone 0.15 mg/kg
Started | 21 | 18 | 21
Completed | 21 | 18 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment Methadone 0.1 mg/kg | Treatment Methadone 0.15 mg/kg | Total
Number analyzed (Participants) | 21 | 18 | 21 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 21 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (13) | 37 (11) | 40 (11) | 40 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 21 | 55
  Male | 3 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 18 | 21 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 9 | 19
  White | 13 | 15 | 12 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 21 | 60
body weight - kg [Mean (Standard Deviation); unit: Kg] | 85 (16) | 88 (42) | 86 (26) | 86 (1.53)
ASA status [Number; unit: units on a scale] — ASA Physical Status Classification System
  ASA I A normal healthy patient Healthy, non-smoking, no or minimal alcohol use ASA II A patient with mild systemic disease without substantive functional limitations.
  ASA III A patient with severe systemic disease with substantive functional limitations;
  units on a scale
    ASA I | 1 | 0 | 0 | 1
    ASA II | 16 | 17 | 21 | 54
    ASA III | 4 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Opioid Administration
Description: Data on opioids administered intraoperatively will be collected from the subject's EMR.
Time Frame: Administered at induction of anesthesia
Measure: Median (Inter-Quartile Range); unit: morphine equivalents mg
Arm/Group | Control | Treatment Methadone 0.1 mg/kg | Treatment Methadone 0.15 mg/kg
Number analyzed (Participants) | 21 | 18 | 21
morphine equivalents mg | 25 [23.3 to 28.3] | 5.6 [5.0 to 6.0] | 8.6 [7.8 to 9.0]
Statistical Analysis 1: Comparison: Control vs Treatment Methadone 0.1 mg/kg vs Treatment Methadone 0.15 mg/kg; Test type: Superiority; p = 0.0001, Chi-squared

2. Primary Outcome: Postoperative Opioid Administration
Description: Data on opioids administered postoperatively will be collected from the subject's EMR. Pain severity will be assessed using Numeric Rating Scale and colored-visual analogue scale. Pain relief postoperatively will be assessed using a 5 point scale [0-no relief, 4-complete relief]
Time Frame: EMR reviewed at 24 hours post-administration or at hospital discharge
Measure: Median (Inter-Quartile Range); unit: morphine equivalents mg
Arm/Group | Control | Treatment Methadone 0.1 mg/kg | Treatment Methadone 0.15 mg/kg
Number analyzed (Participants) | 21 | 18 | 21
morphine equivalents mg | 10 [2.5 to 14.3] | 5.4 [3.3 to 9.6] | 3.3 [0.1 to 5.8]
Statistical Analysis 1: Comparison: Control vs Treatment Methadone 0.1 mg/kg vs Treatment Methadone 0.15 mg/kg; Test type: Superiority; p = 0.01, Kruskal-Wallis

3. Secondary Outcome: Opioid Consumption Within First 30 Postoperative Days
Description: Daily opioid consumption for approx 30 days following surgery (from hospital discharge until postop clinic visit).
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: total postdischarge opioid pills used
Arm/Group | Control | Treatment Methadone 0.1 mg/kg | Treatment Methadone 0.15 mg/kg
Number analyzed (Participants) | 21 | 18 | 21
total postdischarge opioid pills used | 10 [3 to 20] | 7 [4 to 19] | 5 [3 to 13]
Statistical Analysis 1: Comparison: Control vs Treatment Methadone 0.1 mg/kg vs Treatment Methadone 0.15 mg/kg; Test type: Superiority; p = 0.001, Kruskal-Wallis

4. Secondary Outcome: Pain Relief Within First 30 Postoperative Days
Description: Daily pain self-assessments using a numeric (0-10) rating scale were recorded in a home diary for approx 30 days following surgery (from hospital discharge until postop clinic visit). Zero was no pain and 10 was the worst possible pain.
  Patient's 30-day post-discharge scores were averaged individually and compared in between groups.
  In addition, participants recorded pain interference with 7 activities of daily living - mood, ability to walk or move, sleep, normal work outside the home, normal work at home, recreational activities, and enjoyment of life on a 5-point Likert scale. Questions were based on the Patient-Reported Outcomes Measurement Information System Pain Behavior and Pain Interference item banks. Patients also recorded opioid and nonopioid analgesic use, sedation, and time to return to work.
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Treatment Methadone 0.1 mg/kg | Treatment Methadone 0.15 mg/kg
Number analyzed (Participants) | 12 | 14 | 14
score on a scale | 1 [0 to 5] | 1 [0 to 6] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Control vs Treatment Methadone 0.1 mg/kg vs Treatment Methadone 0.15 mg/kg; Test type: Superiority; p = 0.02, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Control | Treatment Methadone 0.1 mg/kg | Treatment Methadone 0.15 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02300077/Prot_SAP_000.pdf